CLINICAL TRIAL: NCT02174640
Title: Acute Effects of Coffee Beverage on Postprandial Inflammation and Oxidative Stress - A Pilot Study
Acronym: COF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-008
Record Dates: First submitted 2014-06-17; First posted 2014-06-25 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Overweight; Obese; Healthy
Keywords: Coffee; Polyphenolics
MeSH Terms: conditions — Overweight; Obesity | interventions — Coffee; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coffee (Active Comparator): Coffee Beverage
  Interventions: Dietary Supplement: Coffee
- Water (Placebo Comparator): Water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Coffee — Coffee Beverage
  Other Names: Active Comparator
  Arms: Coffee
Dietary Supplement: Water — Water
  Other Names: Placebo Comparator
  Arms: Water

SUMMARY:
The primary objective is to test if acute supplementation with Coffee would improve antioxidant status, following consumption of a pro-oxidative high carbohydrate, high fat meal in over weight/ obese humans.

Secondary objective is to determine the ability of coffee to modify postprandial inflammation in overweight/ obese humans.

DETAILED DESCRIPTION:
The proposed study is a single-center, placebo-controlled, randomized, 2-arm, 2-sequence, crossover study that characterize the bioavailability and kinetic profile of coffee over 6-hour postprandial day (PPD).

A planned sample size of 10 will be recruited into the study. This study will require one initial screening visit, pre-study visit, and 2 PPDs. This study will take 3-6 weeks per subject to complete.

The trial will initiate with a screening visit, which will last for about 1-1.5 hours where the subjects' height, weight, waist circumference, fasting blood glucose, fasting hs-CRP (high sensitivity C-reactive protein) concentration, blood pressure and heart rate will be measured and a survey related to general eating, health and exercise habits will be completed.

If willing and eligible to participate, a 3-day food record (2 weekdays and 1 weekend) will be given at the screening visit and collected on the following pre-study Visit to assess subject's baseline dietary intake and pattern. Also, subjects will be instructed to follow a relatively low polyphenolic-diet at least 7 days prior to the first PPD and for the duration of the study. Prior to each PPD, a dinner meal will be provided the day before the PPD to control the second meal effect from food and beverage intake of the night before the PPD.

Subjects will arrive at the center in a fasting state for at least 10 hours, well hydrated and rested. Each PPD will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a registered nurse will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. A standard high carbohydrate and high fat test meal with either 1 cup of coffee or 1 cup of hot water will be served. Thereafter, timers will be started and blood sample will be collected at 20, 40, 60, 120, 180, 240, 300, and 360 minutes for assessment of changes in inflammation markers and relative metabolic indices. The sequence of receiving the coffee or hot water treatment at each visit will be randomly assigned based on computer generated sequences: hot water- coffee or coffee-hot water.

Premenopausal female subjects will be studied during the follicular phase of their menstrual cycle because food intake tends to be more stable during the follicular phase (days 1-13) than during the luteal phase (days 14-28) when the rise in progesterone levels decrease satiety and often resulting in increased intake. Both PPD visits will be placed at least 3 days apart as well.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with regular menstrual cycle
* Aged between 20 to 45 years old
* Body Mass Index (BMI) range from 25 to 35 kg/m2; exception BMI 23 to 35 kg/m2 for Asian population
* Fasting blood glucose concentration < 110 mg/dL
* Fasting hs-CRP >2 mg/dL to < 10 mg/dL
* Weight stable: not gained or lost weight +/- 5 lbs in previous 3 months
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications or dietary supplements that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, fish oil, probiotics, grape seed supplement, etc…If anti-inflammation and/or antibiotic medications/supplements are taken, subjects may qualify if go off these medications/supplements 30 days wash-out before entering the study.
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol

Exclusion Criteria:

* Men
* Past smokers: abstinence for less than 2 years
* Women who smoke
* Women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compound or any their stated ingredients.
* Women known to have/diagnosed with diabetes mellitus
* Women who have fasting blood glucose concentrations ≥110 mg/dL
* Women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries.
* Women with cancer other than non-melanoma skin cancer in previous 5 years.
* Women who are taking medication or dietary supplements that may interfere with the outcomes of the study; e.g., antioxidant supplements, anti-inflammation, lipid lowering medication. Subjects may choose to go off dietary supplements (requires 30 days washout).
* Women who are taking blood pressure lowering medication that may interfere with the outcomes of the study; e.g. diuretics.
* Women who have donated blood within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Women who are vegetarians or vegans
* Substance (alcohol or drug) abuse within the last 2 years.
* Excessive coffee and tea consumers (> 4 cups/day); berry and grape consumers (>2 cups/day)
* Women who do excessive exercise regularly or athlete
* Unstable weight: gained or lost weight +/- 5 lbs in previous 3 months
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06-15 (Actual); Primary Completion 2014-10-27 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
Changes in plasma inflammation markers over 6 hours after coffee or hot water consumption with a high carbohydrate and high fat meal. | 6 hours
  The influence of coffee consumption on inflammation markers

SECONDARY OUTCOMES:
Changes in plasma metabolic markers over 6 hours after coffee or hot water consumption with a high carbohydrate and high fat meal | 6 hours
  The influence of coffee consumption on metabolic markers

OTHER OUTCOMES:
Changes in oxidative stress markers over 6 hours after coffee or hot water consumption with a high carbohydrate and high fat meal | 6 hours
  The influence of coffee consumption on oxidative stress markers

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No